CLINICAL TRIAL: NCT06404684
Title: Paraphilic Disorders and Other Conditions With Risk for Sexual Violence: the Evaluation of an Adapted Cognitive Behavioral Therapy (CBT) Manual for Paraphilic Disorders
Brief Title: Psychological Treatment for Paraphilic Disorders
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Josephine Savard, Principal Investigator, Region Stockholm
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-01882-02
Record Dates: First submitted 2024-04-30; First posted 2024-05-08 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Paraphilic Disorders
Keywords: paraphilic disorders
MeSH Terms: conditions — Paraphilic Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: we will use a multiple baseline single-case experimental design (SCED) with phase A (baseline) and phase B (treatment).
  Participants are randomized to different lengths of phase A; 15-21 days, so-called open randomization.
  Phase B is the CBT treatment. The B phase aims to last 84 days (12 weeks).
  Seven participants will be included with the main diagnosis of voyeurism, exhibitionism and/or frotteurism, and seven participants with coercive-sexual sadism disorder. The participants in each group will be randomized to seven lengths of phase A. These two groups of seven participants will be treated and analyzed separately.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cognitive behavioral therapy (CBT) (Experimental): The current CBT-manual is based on the CBT-manual used for hypersexual disorder, which was developed by ANOVA and evaluated scientifically, (Hallberg 2017, 2019, 2020), but has now been adapted to better meet the current target group. The CBT manual addresses specific sexual problematic behaviors but also contains interventions to deal with comorbidity (e.g. depression and anxiety). The treatment consists of 10 modules and is given by a psychologist (face to face or video).
  Interventions: Behavioral: Cognitive behavioral therapy (CBT)

INTERVENTIONS:
Behavioral: Cognitive behavioral therapy (CBT) — se above

SUMMARY:
The goal of this randomized study is to learn if a psychological intervention can treat help-seeking patients with paraphilic disorders.

The main questions it aims to answer are:

1. Is psychological therapy helpful for the reduction of problematic sexual behaviors among patients with paraphilic disorders?
2. Is psychological helpful for the reduction of psychiatric symptoms and risk factors for sexual violence and improving quality of life among patients with paraphilic disorders?
3. How do patients with paraphilic disorders describe pathways to care (e.g. perceived obstacles to seeking care) and how do they experience the treatment?

The treatment addresses specific sexual problems. It also addresses mental symptoms (e.g. depression and anxiety). A psychologist provides the treatment face to face (on site or video). The aim is to finish the treatment within 12 weeks.

The patient will report symptoms on a daily basis. The patient will also be interviewed after completion of treatment. The investigator will pose questions such as "Was there anything that was experienced as particularly helpful in the treatment?", "Was there anything that was not helpful?". The investigator will also ask about treatment seeking behavior with questions such as "What kinds of resources would be helpful if they were available?"

DETAILED DESCRIPTION:
The aim with this study is to systematically evaluate Cognitive Behavioral Therapy (CBT) for help-seeking patients with paraphilic disorders. The CBT-manual that will be used has been adapted to meet the current target group. The investigators will also interview the participants on how they experience the treatment and their pathways to care (e.g., perceived obstacles to seeking care).

1. Is CBT effective for the reduction of problematic sexual behaviors among individuals with paraphilic disorders?
2. Is CBT effective for the reduction of psychiatric comorbidity and risk factors for sexual violence and improving quality of life among individuals with paraphilic disorders?
3. How do men with paraphilic disorders describe pathways to care (e.g., perceived obstacles to seeking care) and how do they experience the CBT treatment?

To answer questions a-b, the investigators will use a multiple baseline single-case experimental design (SCED) with phase A (baseline) and phase B (treatment). The participants will answer four questions daily, and additional questionnaires before phase A, before phase B, middle of phase B and at end of treatment.

Primary endpoint is the last reported measurement in phase B. The investigators will also have a follow-up measurement after 3 months.

To answer question c, qualitative interviews about perceived effect of treatment will be conducted. The interviews will transcribed and analyzed. The participants will also answer questionnaires addressing expectancy, perceived satisfaction, and negative effect of treatment.

Overall, a mixed method will be used to answer all three questions.

Procedures Patients seeking treatment at ANOVA (Karolinska University Hospital, Sweden) who is included in Paraphilic Disorders and Other Conditions With Risk for Sexual Violence: a Case-control Study (ClinicalTrials.gov identifier NCT05861752, please see the detailed description for an explanation of study procedures including assessments), and meet the inclusion/exclusion criteria below will be included in this project.

Seven participants will be included with the main diagnosis of voyeurism, exhibitionism and/or frotteurism, and seven participants with coercive-sexual sadism disorder. These two groups of seven participants will be treated and analyzed separately.

Termination criteria

1. Conditions that are deemed to complicate the treatment (e.g., drug abuse or the development of a serious mental disorder).
2. The treatment is deemed insufficient to meet the patient's needs.

Analytical plan SCED is useful to evaluate a new/adapted treatment where the conditions being studied are rare, and/or the group being studied is heterogeneous (Krasny-Pacini & Evans, 2018).

A traditional power analysis is not feasible in SCED. Instead, power is achieved through repeated measurements. It has been recommended to include at least 3 participants, at least 3 (preferably 5) measurements per person at baseline, or at least three measurable behaviors. Moreover, randomization to at least 3 different lengths of the baseline phase has been suggested (Krasny-Pacini & Evans, 2018) while others advocate at least 6 (Kratochwill et al., 2013).

Therefore, 7 participants will be randomized to 7 lengths of the baseline phase. Three different problematic sexual behaviors will be assessed daily (main outcome).

The data will be analyzed visually and descriptively to see changes in different phases: level lines (mean/median value), trends, variability, immediacy of effect and consistency (Kratochwill et al., 2013).

Kendal's Tau/Tau U will be used to analyze statistical differences in the variables between the phases.

Effect size on the outcome measures will be reported as standardized mean value.

Missing data will be handled by using the average of neighboring data points. Other outcome measures will be examined and reported descriptively and as percentage improvement.

ELIGIBILITY:
Inclusion Criteria:

1. Participants included in the study Paraphilic Disorders and Other Conditions With Risk for Sexual Violence: a Case-control Study
2. Deemed to benefit from CBT.
3. Signed informed consent form for participation in the CBT treatment.

Exclusion Criteria:

1. Mental condition that could negatively influence either the patient's health or the scientific aspects of the study, e.g., substance use syndrome, other ongoing psychotherapeutic treatment.
2. Initiation of medication or change change of concurrent medication or dosage in the past three months regarding antidepressants, attention deficit hyperactivity disorder medication, cortisone, testosterone, naltrexone, testosterone blockers, or dopamine precursors. Smaller adjustments may in some cases be acceptable (assessed by study psychiatrist).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2025-03-04 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Questions about sexual behaviors ("diary") | From date of randomization until the date of end of treatment (week 12), and a follow-up assessement 3 months after end of treatment.
  Three questions about time spent on problematic sexual behaviors or fantasies, level of desire and sex as coping.
  Each question is scored 0-4. The main outcome measure is the total score of these three questions (0-12 points). A higher score indicates more severe problems.
Questions about sexual behaviors ("diary") | From date of randomization until the date of end of treatment (week 12), and a follow-up assessement 3 months after end of treatment.
  Three questions about time spent on problematic sexual behaviors or fantasies, level of desire and sex as coping.
  Each question is scored 0-4. The three problem areas described under main outcome are handled as separate items and analyzed separately. A higher score indicates more severe problems.
Frotteuristic Disorder:Current Assessment Scale (FD: CAS) | start of randomization (phase A), start of treatment (phase B), in the middle of treatment (week 6), at end of treatment (week 12), and follow-up 3 months after treatment.
  The questionnaire will be used if the participant has a diagnosis of frotteuristic disorder. The questionnaire assesses frotteuristic behaviors. The questionnaire is scored 0-32. A higher score indicates more severe problems.
Voyeuristic Disorder: Current Assessment Scale (VD: CAS) | start of randomization (phase A), start of treatment (phase B), in the middle of treatment (week 6), at end of treatment (week 12), and follow-up 3 months after treatment.
  The questionnaire will be used if the participant has a diagnosis of voyeuristic disorder. The questionnaire assesses voyeuristic behaviors. The questionnaire is scored 0-32. A higher score indicates more severe problems.
Exhibitionistic Disorder: Current Assessment Scale (ED: CAS), | start of randomization (phase A), start of treatment (phase B), in the middle of treatment (week 6), at end of treatment (week 12), and follow-up 3 months after treatment.
  The questionnaire will be used if the participant has a diagnosis of exhibitionistic disorder. The questionnaire assesses exhibitionistic behaviors. The questionnaire is scored 0-32. A higher score indicates more severe problems.
Coercive Sexual Sadism Disorder: Current Assessment Scale (CSSD: CAS) | start of randomization (phase A), start of treatment (phase B), in the middle of treatment (week 6), at end of treatment (week 12), and follow-up 3 months after treatment.
  The questionnaire will be used if the participant has a diagnosis of Coercive Sexual Sadism Disorder. The questionnaire assesses coercive and sadistic (sexual) behaviors. The questionnaire is scored 0-32. A higher score indicates more severe problems.

SECONDARY OUTCOMES:
A question about general well-being | From date of randomization until the date of end of treatment (week 12), and a follow-up assessement 3 months after end of treatment.
  A question from general well-being schedule, scored 0-6. A higher score indicates more severe problems.
Hospital Anxiety and Depression Scale (HADS) | start of randomization (phase A), start of treatment (phase B), in the middle of treatment (week 6), at end of treatment (week 12), and follow-up 3 months after treatment.
  Score range is 0-21. A higher score indicates more severe problems.
The Brief version of the Difficulties in emotional regulation scale (DERS-16) | start of randomization (phase A), start of treatment (phase B), in the middle of treatment (week 6), at end of treatment (week 12), and follow-up 3 months after treatment.
  Score range is 16-80. A higher score indicates more severe problems.
Brunnsviken Brief Quality of Life Inventory (BBQ) | start of randomization (phase A), start of treatment (phase B), in the middle of treatment (week 6), at end of treatment (week 12), and follow-up 3 months after treatment.
  Score range is 0-48. A higher score indicates high quality of life
Perceived Social Support (PSS-14) | start of randomization (phase A), start of treatment (phase B), in the middle of treatment (week 6), at end of treatment (week 12), and follow-up 3 months after treatment.
  Two subscales, one addressing support from family and the other from friends. Score range is 20-80. A higher score indicates more severe problems.
Revised University of California, Los Angeles (UCLA) Loneliness Scale (RULS) | start of randomization (phase A), start of treatment (phase B), in the middle of treatment (week 6), at end of treatment (week 12), and follow-up 3 months after treatment.
  Score range is 20-80. A higher score indicates more loneliness.
the rape questionnaire | start of randomization (phase A), start of treatment (phase B), in the middle of treatment (week 6), at end of treatment (week 12), and follow-up 3 months after treatment.
  Assessment of cognitive distortions about sex. Score range is 36-144. A higher score indicate more severe problems.
Hypersexual Behavior Inventory (HBI) | start of randomization (phase A), start of treatment (phase B), in the middle of treatment (week 6), at end of treatment (week 12), and follow-up 3 months after treatment.
  a 19-item scale constructed to reflect the proposed Diagnostic and statistical manual of mental disorders, 5th edition criteria of hypersexual disorder. Score range is 19-95. A higher score indicates more severe problems.
Credibility/Expectancy questionnaire (CEQ) | Before treatment starts
  Two subscales with questions about treatment credibility and treatment outcome expectations. Four questions are rated on a scale of 1 to 9 (not at all to a lot), 2 questions are rated from 0% to 100%. A higher score indicate more credibility and expectancy.
Negative effect of treatment (NEQ) | After completion of treatment (week 12)
  It contains 32 items that are scored on a five point Likert-scale (0-4) and differentiates between negative effects that are attributed to treatment and those possibly caused by other circumstances, as well as one open-ended question.
Client Satisfaction Scale-8 (CSQ-8) | After completion of treatment (week 12)
  Score range is 8-32. A higher score indicates higher treatment satisfaction

OTHER OUTCOMES:
Qualitative interview (research question c) | After completion of treatment (week 12)
  A 60 min interview questions such as "Can you tell us about the treatment you received", "What do you take with you from the treatment?", "Was there anything that you experienced as particularly helpful in the treatment?", "Was there anything that was not helpful?"
Quality assurance of the manual after each module | After each treatment module (i.e., 10 times under a time-period of 12 weeks)
  Include questions such as "how relevant and helpful did you find the current module on a scale of 1-5 (1 = not at all helpful, 3 = neither, 5 = very helpful), How much time did you spend working on the material (reading and doing homework)?

CONTACTS AND LOCATIONS:
Overall Officials: josephine Savard, Principal Investigator — Anova, Karolinska University Hospital, Stockholm, Sweden
Locations (1):
- ANOVA, Karolinska university hospital, Stockholm, Stockholm County, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Individual participants' data that underlie the results of the published article, after deidentification (text, tables, figures and appendices) might be available to researches who provide a methodically sound proposal.
Supporting Information: Study Protocol, ICF
Time Frame: Immediately following publication and ending ten years from study completion.
Access Criteria: Researches who provide a methodically sound proposal. Proposals should be directed to the PI. To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Background] Kratochwill TR, Horner RH, Levin JR, Machalicek W, Ferron J, Johnson A. Single-case intervention research design standards: Additional proposed upgrades and future directions. J Sch Psychol. 2023 Apr;97:192-216. doi: 10.1016/j.jsp.2022.12.002. Epub 2023 Feb 22. PMID 36914365
- [Background] Krasny-Pacini A, Evans J. Single-case experimental designs to assess intervention effectiveness in rehabilitation: A practical guide. Ann Phys Rehabil Med. 2018 May;61(3):164-179. doi: 10.1016/j.rehab.2017.12.002. Epub 2017 Dec 15. PMID 29253607
- [Background] Hallberg J, Kaldo V, Arver S, Dhejne C, Piwowar M, Jokinen J, Oberg KG. Internet-Administered Cognitive Behavioral Therapy for Hypersexual Disorder, With or Without Paraphilia(s) or Paraphilic Disorder(s) in Men: A Pilot Study. J Sex Med. 2020 Oct;17(10):2039-2054. doi: 10.1016/j.jsxm.2020.07.018. Epub 2020 Sep 6. PMID 32900671
- [Background] Hallberg J, Kaldo V, Arver S, Dhejne C, Oberg KG. A Cognitive-Behavioral Therapy Group Intervention for Hypersexual Disorder: A Feasibility Study. J Sex Med. 2017 Jul;14(7):950-958. doi: 10.1016/j.jsxm.2017.05.004. Epub 2017 Jun 8. PMID 28602666
- [Background] Hallberg J, Kaldo V, Arver S, Dhejne C, Jokinen J, Oberg KG. A Randomized Controlled Study of Group-Administered Cognitive Behavioral Therapy for Hypersexual Disorder in Men. J Sex Med. 2019 May;16(5):733-745. doi: 10.1016/j.jsxm.2019.03.005. Epub 2019 Apr 5. PMID 30956109